CLINICAL TRIAL: NCT02759315
Title: A Phase II, Open-Label Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-3682 + MK-8408 in Subjects With Chronic HCV Genotype 1, 2, 3, 4, 5 or 6 Infection
Brief Title: Efficacy and Safety of Uprifosbuvir (MK-3682) With Ruzasvir (MK-8408) in Adults With Chronic Hepatitis C Genotype 1, 2, 3, 4, 5 or 6 Infection (MK-3682-035)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated based on review of Phase 2 efficacy data
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3682-035; MK-3682-035 (Other: Merck Registration Number)
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — uprifosbuvir; ruzasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- GT1: Uprifosbuvir 450 mg + Ruzasvir 60 mg (Experimental): Participants will receive an oral dose of 450 mg uprifosbuvir (3 x 150 mg tablets) and 60 mg ruzasvir (6 x 10 mg capsules) following an overnight fast and at least one hour before a meal, once a day, for 12 weeks. The GT1 Arm is sub-divided into GT1a and GT1b Arms. GT1a Arm will enroll approximately 35 participants including up to 10 participants who are compensated cirrhotics and GT1b Arm will enroll approximately 15 participants including up to 5 participants who are compensated cirrhotics.
  Interventions: Drug: Uprifosbuvir 450 mg; Drug: Ruzasvir 60 mg
- GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg (Experimental): Participants will receive an oral dose of 450 mg uprifosbuvir (3 x 150 mg tablets) and 60 mg ruzasvir (6 x 10 mg capsules) following an overnight fast and at least one hour before a meal, once a day, for 12 weeks. The GT2 Arm of the study will enroll approximately 50 participants including up to 15 participants who are compensated cirrhotics.
  Interventions: Drug: Uprifosbuvir 450 mg; Drug: Ruzasvir 60 mg
- GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg (Experimental): Participants will receive an oral dose of 450 mg uprifosbuvir (3 x 150 mg tablets) and 60 mg ruzasvir (6 x 10 mg capsules) following an overnight fast and at least one hour before a meal, once a day, for 12 weeks. The GT3 Arm of the study will enroll approximately 50 participants including up to 15 participants who are compensated cirrhotics.
  Interventions: Drug: Uprifosbuvir 450 mg; Drug: Ruzasvir 60 mg
- GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg (Experimental): Participants will receive an oral dose of 450 mg uprifosbuvir (3 x 150 mg tablets) and 60 mg ruzasvir (6 x 10 mg capsules) following an overnight fast and at least one hour before a meal, once a day, for 12 weeks. The GT4 Arm of the study will enroll approximately 50 participants including up to 15 participants who are compensated cirrhotics.
  Interventions: Drug: Uprifosbuvir 450 mg; Drug: Ruzasvir 60 mg
- GT5: Uprifosbuvir 450 mg + Ruzasvir 60 mg (Experimental): Participants will receive an oral dose of 450 mg uprifosbuvir (3 x 150 mg tablets) and 60 mg ruzasvir (6 x 10 mg capsules) following an overnight fast and at least one hour before a meal, once a day, for 12 weeks. The GT5 Arm of the study will enroll approximately 25 participants including both non- cirrhotics and compensated cirrhotics.
  Interventions: Drug: Uprifosbuvir 450 mg; Drug: Ruzasvir 60 mg
- GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg (Experimental): Participants will receive an oral dose of 450 mg uprifosbuvir (3 x 150 mg tablets) and 60 mg ruzasvir (6 x 10 mg capsules) following an overnight fast and at least one hour before a meal, once a day, for 12 weeks. The GT6 Arm of the study will enroll approximately 25 participants including both non- cirrhotics and compensated cirrhotics.
  Interventions: Drug: Uprifosbuvir 450 mg; Drug: Ruzasvir 60 mg

INTERVENTIONS:
Drug: Uprifosbuvir 450 mg — 450 mg administered as 3 x 150 mg oral tablets
  Other Names: MK-3682
Drug: Ruzasvir 60 mg — 60 mg administered as 6 x 10 mg oral capsules
  Other Names: MK-8408

SUMMARY:
This study is an open-label, multi-center trial to evaluate the novel 2-drug regimen of uprifosbuvir (MK-3682) 450 mg and ruzasvir (MK-8408) 60 mg in participants with chronic hepatitis C virus (HCV) genotype (GT)1, GT2, GT3, GT4, GT5, or GT6 infection. The impact of the study treatment regimen on the percentage of participants with undetectable HCV ribonucleic acid [RNA] 12 weeks after completing study treatment (SVR12) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Has hepatitis C virus (HCV) ribonucleic acid (RNA) at the time of screening
* Has documented chronic HCV genotype (GT)1, GT2, GT3, GT4, GT5, or GT6 with no evidence of non-typeable or mixed GT infection
* Is otherwise healthy as determined by the medical history, physical examination, electrocardiogram (ECG), and clinical laboratory measurements performed at the time of screening
* Has absence of cirrhosis or has compensated cirrhosis
* Is HCV treatment-naïve or has experienced virologic failure after completing a prior interferon-containing regimen
* Is of non-childbearing potential or agrees to avoid becoming pregnant or impregnating a partner beginning at least 2 weeks prior to administration of the initial dose of study drug and for 14 days after the last dose of study drug
* For human immunodeficiency virus (HIV) co-infected participants: is not currently on antiretroviral therapy (ART) and has no plans to initiate ART treatment while participating in this study Or has well-controlled HIV on ART

Exclusion Criteria:

* Is mentally or legally incapacitated, has significant emotional problems (at screening or expected during the study) or has a history of a clinically significant psychiatric disorder that would interfere with the study procedures.
* Has evidence of decompensated liver disease manifested by the presence of or history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver disease
* Is Child-Pugh Class B or C or has a Pugh-Turcotte (CPT) score >6 if cirrhotic
* Is co-infected with Hepatitis B Virus
* Has a history of opportunistic infection in the preceding 6 months prior to screening if co-infected with HIV
* Has a history of malignancy ≤5 years prior to study start (except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or carcinoma in situ) or is under evaluation for other active or suspected malignancy
* Has cirrhosis and liver imaging within 6 months prior to study start showing evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC
* Is taking any medications or herbal supplements restricted by the study entry criteria in the period from ≤2 weeks prior to study start through 2 weeks after the last dose of study drug
* Has clinically-relevant drug or alcohol abuse within 12 months of study start
* Has participated in any clinical study of an investigational product within 30 days prior to the first dose of study drug
* Is female and is pregnant or breastfeeding, or expecting to conceive or donate eggs from at least 2 weeks prior to study start and 14 days after the last dose of study drug
* Is male and is expecting to donate sperm from at least 2 weeks prior to Day 1 until 14 days after the last dose of study drug
* Has or has had any of the following: organ transplants (including hematopoietic stem cell transplants) other than cornea and hair; poor venous access; history of gastric surgery; or history of malabsorption disorders
* Has any cardiac abnormalities/dysfunction including but not limited to: unstable angina; unstable congestive heart failure; or unstable arrhythmia
* Has a history of a medical/surgical condition that resulted in hospitalization within 3 months prior to study start, other than for minor elective procedures
* Has any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids, tumor necrosis factor (TNF) antagonists, or other immunosuppressant drugs during the study
* Has evidence of history of chronic hepatitis not caused by HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lawitz E, Poordad F, Anderson LJ, Vesay M, Kelly MM, Liu H, Gao W, Fernsler D, Asante-Appiah E, Robertson MN, Hanna GJ, Barr E, Butterton J, Kowdley KV, Hassanein T, Sahota A, Gordon SC, Yeh WW. Efficacy and safety of ruzasvir 60 mg and uprifosbuvir 450 mg for 12 weeks in adults with chronic hepatitis C virus genotype 1, 2, 3, 4 or 6 infection. J Viral Hepat. 2019 Jun;26(6):675-684. doi: 10.1111/jvh.13079. Epub 2019 Mar 12. PMID 30739366
- [Derived] Lawitz E, Gane E, Feld JJ, Buti M, Foster GR, Rabinovitz M, Burnevich E, Katchman H, Tomasiewicz K, Lahser F, Jackson B, Shaughnessy M, Klopfer S, Yeh WW, Robertson MN, Hanna GJ, Barr E, Platt HL; C-BREEZE-2 Study Investigators. Efficacy and safety of a two-drug direct-acting antiviral agent regimen ruzasvir 180 mg and uprifosbuvir 450 mg for 12 weeks in adults with chronic hepatitis C virus genotype 1, 2, 3, 4, 5 or 6. J Viral Hepat. 2019 Sep;26(9):1127-1138. doi: 10.1111/jvh.13132. Epub 2019 Jul 11. PMID 31108015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with hepatitis C virus (HCV) genotype (GT) 1, 2, 3, 4, or 6 infection were enrolled at 5 study centers in the United States. Participants with HCV GT5 infection were initially intended for inclusion but none were enrolled.
Groups:
- GT1: Uprifosbuvir 450 mg + Ruzasvir 60 mg: Participants with HCV GT1 infection took uprifosbuvir 450 mg ruzasvir 60 mg once daily for 12 weeks. Study drug was taken after an overnight fast and at least 1 hour before a meal.
- GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg: Participants with HCV GT2 infection took uprifosbuvir 450 mg ruzasvir 60 mg once daily for 12 weeks. Study drug was taken after an overnight fast and at least 1 hour before a meal.
- GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg: Participants with HCV GT3 infection took uprifosbuvir 450 mg ruzasvir 60 mg once daily for 12 weeks. Study drug was taken after an overnight fast and at least 1 hour before a meal.
- GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg: Participants with HCV GT4 infection took uprifosbuvir 450 mg ruzasvir 60 mg once daily for 12 weeks. Study drug was taken after an overnight fast and at least 1 hour before a meal.
- GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg: Participants with HCV GT6 infection took uprifosbuvir 450 mg ruzasvir 60 mg once daily for 12 weeks. Study drug was taken after an overnight fast and at least 1 hour before a meal.
Period: Overall Study
Arm/Group | GT1: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg
Started | 69 | 29 | 39 | 20 | 3
Completed | 65 | 28 | 29 | 19 | 2
Not Completed | 4 | 1 | 10 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 4 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Study terminated prior to completion | 2 | 0 | 5 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GT1: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg | Total
Number analyzed (Participants) | 69 | 29 | 39 | 20 | 3 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (10.7) | 57.2 (6.8) | 48.7 (10.3) | 56.5 (8.5) | 61.3 (1.5) | 51.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 10 | 18 | 5 | 1 | 67
  Male | 36 | 19 | 21 | 15 | 2 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 0 | 1 | 0 | 7
  White | 64 | 27 | 39 | 19 | 0 | 149
  More than one race | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks After Completing Study Therapy (SVR12)
Description: The percentage of participants in each arm achieving SVR12 was determined. SVR12 was defined as HCV ribonucleic acid (RNA) levels in plasma < lower limit of quantification (LLOQ) 12 weeks after completing study treatment. Plasma levels of HCV RNA were measured with the COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0 ® assay, which has a LLOQ of 15 IU/mL.
Time Frame: Week 24 (12 weeks after completing study therapy)
Population: All participants who received ≥1 dose of study treatment, have data available, who do not have protocol deviations that could substantially affect the results of the endpoint, and who did not discontinue from the study for non-treatment-related reasons, are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | GT1: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg
Number analyzed (Participants) | 69 | 28 | 39 | 20 | 3
Percentage of Participants | 97.1 [89.9 to 99.6] | 100.0 [87.7 to 100.0] | 76.9 [60.7 to 88.9] | 90.0 [68.3 to 98.8] | 66.7 [9.4 to 99.2]

2. Primary Outcome: Percentage of Participants With ≥1 Adverse Events (AEs)
Description: The percentage of participants experiencing an AE during the treatment period and first 2 weeks of follow-up was determined. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to Week 14 (up to 2 weeks after completing study therapy)
Population: All participants who received ≥1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | GT1: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg
Number analyzed (Participants) | 69 | 29 | 39 | 20 | 3
Percentage of Participants | 52.2 | 44.8 | 43.6 | 55.0 | 66.7

3. Primary Outcome: Percentage of Participants Withdrawing From Study Therapy Due to an AE
Description: The percentage of participants discontinuing from study therapy during the treatment period was determined. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to Week 12
Population: All participants who received ≥1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | GT1: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg
Number analyzed (Participants) | 69 | 29 | 39 | 20 | 3
Percentage of Participants | 0.0 | 3.4 | 0.0 | 5.0 | 0.0

4. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks After Completing Study Therapy (SVR24)
Description: The percentage of participants in each arm achieving SVR24 was determined. SVR24 was defined as HCV RNA levels in plasma < LLOQ 24 weeks after completing study treatment. Plasma levels of HCV RNA were measured with the COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0 ® assay, which has a LLOQ of 15 IU/mL. For SVR24, participants with GT1 infection were separated into GT1a or GT1b infection.
Time Frame: Week 36 (24 weeks after completing study therapy)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Groups:
- GT1a: Uprifosbuvir 450 mg + Ruzasvir 60 mg: Participants with HCV GT1a infection took uprifosbuvir 450 mg ruzasvir 60 mg once daily for 12 weeks. Study drug was taken after an overnight fast and at least 1 hour before a meal.
- GT1b: Uprifosbuvir 450 mg + Ruzasvir 60 mg: Participants with HCV GT1b infection took uprifosbuvir 450 mg ruzasvir 60 mg once daily for 12 weeks. Study drug was taken after an overnight fast and at least 1 hour before a meal.
Arm/Group | GT1a: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT1b: Uprifosbuvir 450 mg + Ruzasvir 60 mg
Number analyzed (Participants) | 53 | 28 | 36 | 20 | 3 | 14
Percentage of Participants | 96.2 | 100.0 | 75.0 | 90.0 | 66.7 | 100.0

5. Secondary Outcome: Percentage of Participants With Virologic Failure (VF)
Description: The percentage of participants in each arm experiencing VF was determined. VF was defined as: 1) non-response (HCV RNA detected at end of treatment without HCV RNA < LLOQ while on treatment); 2) rebound (>1 log 10 IU/mL increase in HCV RNA from nadir while on treatment); 3) virologic breakthrough (HCV RNA ≥LLOQ after being <LLOQ on treatment); or 4) relapse (HCV RNA ≥LLOQ after end of all study therapy after being undetectable at end of treatment); virologic failure could occur either on-treatment or relapse post-treatment. For VF, participants with GT1 infection were separated into GT1a or GT1b infection
Time Frame: 12 weeks after the end of all study therapy (24 weeks)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | GT1a: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT1b: Uprifosbuvir 450 mg + Ruzasvir 60 mg
Number analyzed (Participants) | 54 | 28 | 39 | 20 | 3 | 15
Percentage of Participants | 3.7 | 0.0 | 23.1 | 5.0 | 33.3 | 0.0

6. Secondary Outcome: Percentage of Participants With Baseline Resistance-Associated Substitutions (RAS) Achieving SVR12
Description: The percentage of participants in each arm with baseline RAS achieving SVR12 was determined. Analysis of RAS in NS5A or NS5B at baseline was determined. SVR12 was defined as HCV RNA levels in plasma < LLOQ 24 weeks after completing study treatment. Plasma levels of HCV RNA were measured with the COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0 ® assay, which has a LLOQ of 15 IU/mL.
Time Frame: 12 weeks after the end of all study therapy (24 weeks)
Population: All participants who received ≥1 dose of study treatment, and who do not have protocol deviations that could substantially affect the results of the endpoint, and who did not discontinue from the study for non-treatment-related reasons, and who had baseline sequencing data available, are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | GT1: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg
Number analyzed (Participants) | 69 | 28 | 39 | 19 | 3
Percentage of Participants | 97.1 | 100.0 | 97.4 | 94.7 | 66.6

7. Primary Outcome: Percentage of Participants With ≥1 Events of Clinical Interest (ECIs)
Description: The percentage of participants with ECIs was determined. ECIs were defined as the following: 1) an overdose of study drug; 2) first instance of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >500 IU/L; 3) first instance of ALT or AST >3x nadir and >3x upper limit of normal (ULN); 4) first instance of estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m^2; or 4) first instance of serum creatinine >1.3x ULN and elevated from baseline.
Time Frame: Up to Week 14 (up to 2 weeks after completing study therapy)
Population: All participants who received ≥1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | GT1: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg
Number analyzed (Participants) | 69 | 29 | 39 | 20 | 3
Percentage of Participants
  Overdose: number analyzed (Participants) | 3 | 1 | 2 | 0 | 0
  Overdose | 4.3 | 3.4 | 5.1 |  |
  Non-overdose ECI: number analyzed (Participants) | 2 | 0 | 1 | 0 | 0
  Non-overdose ECI | 2.8 |  | 2.5 |  |

ADVERSE EVENTS:
Time Frame: Up to 36 weeks (up to 24 weeks after completing study treatment)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. All participants who received ≥1 dose of study drug are included.
Arm/Group | GT1: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg | GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/29 | 1/39 | 0/20 | 0/3
Serious Adverse Events (participants affected / at risk) | 4/69 | 0/29 | 1/39 | 2/20 | 0/3
Other Adverse Events (participants affected / at risk) | 25/69 | 8/29 | 13/39 | 6/20 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GT1: Uprifosbuvir 450 mg + Ruzasvir 60 mg (N=69) | GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg (N=29) | GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg (N=39) | GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg (N=20) | GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg (N=3)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GT1: Uprifosbuvir 450 mg + Ruzasvir 60 mg (N=69) | GT2: Uprifosbuvir 450 mg + Ruzasvir 60 mg (N=29) | GT3: Uprifosbuvir 450 mg + Ruzasvir 60 mg (N=39) | GT4: Uprifosbuvir 450 mg + Ruzasvir 60 mg (N=20) | GT6: Uprifosbuvir 450 mg + Ruzasvir 60 mg (N=3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Fatigue (General disorders) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT02759315/Prot_SAP_000.pdf